CLINICAL TRIAL: NCT00276900
Title: Prevention of Recurrent Postpartum Depression
Brief Title: Sertraline for the Prevention of Recurrent Postpartum Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Wisner, Professor of Psychiatry, Obstetrics and Gynecology and Reproductive Sciences, Epidemiology and Women's Studies, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH053735 (NIH); R01MH053735 (NIH); DSIR 83-ATP
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Depression
Keywords: Postpartum Depression; Recurrent Depression
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sertraline

SUMMARY:
This study will determine the effectiveness of taking sertraline within 24 hours of giving birth in preventing a recurrence of postpartum depression.

DETAILED DESCRIPTION:
Depression after pregnancy is called postpartum depression and may be caused by a rapid change in hormone levels during and immediately after pregnancy. Researchers believe that it is one of the most common complications linked to pregnancy. This type of depression occurs in 10 to 15% of women within the first 3 months of giving birth and it can negatively affect both mothers and their children. Mothers with postpartum depression may experience low energy, difficulty concentrating, irritability, and inability to meet their children's needs for love and affection. Research shows that children of mothers with postpartum depression may have delays in language development, difficulty with emotional bonding to others, behavioral problems, lower activity levels, sleep problems, and distress. Many women who have suffered from postpartum depression in the past are worried about a repeat episode with the birth of their next baby. This study will determine the effectiveness of taking sertraline within 24 hours of giving birth in preventing a recurrence of postpartum depression.

Participants in this double blind study will initially report to the study site two separate times while they are pregnant. At the first visit, which will last approximately 3 hours, medical and psychiatric histories will be taken. Blood and urine samples will also be collected at this time. At the second visit, which will last approximately 1 hour, participants will be randomly assigned to receive either sertraline or placebo for the year following childbirth. All participants will then either attend 10 clinic visits, each lasting 1 hour, or receive 17 phone calls over the course of the first 28 weeks postpartum. Mood symptoms and day-to-day functioning will be assessed. If the participant's baby is being breastfed, a blood sample will also be taken from the baby at Week 4 postpartum. At Week 12 postpartum, the baby will wear an actigraph to measure his or her activity for one week. At Week 24 postpartum, participants who are not depressed will be randomly assigned to either continue on sertraline or taper to placebo over 4 weeks. Those who were originally assigned to receive placebo will continue taking placebo for the remainder of the study. Starting at Week 29 postpartum, there will be approximately one clinic visit per month for the remainder of the year. Participants' functioning, ability to interact with their children, and symptoms of depression will be assessed at these visits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Presents by week 36 gestation for first two study visit interviews (interviews may be combined)
* History of DSM-IV Major Depression after the age of 15
* Score no higher than 19 on the 29-item SIGH-ADS at Week 36
* Medically healthy, as determined by a physician

Exclusion criteria

* Current major depression
* Urine screen positive for drugs
* Currently using other therapies for depression
* DSM-IV diagnoses of bipolar 1 or 2 disorder or any psychotic episode
* History of substance abuse within 6 months prior to study entry
* Has not received any obstetrical care
* Use of medications for medical disorders (except for treatment of stable disorders)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2003-12; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms (measured at Weeks 24 and 52 postpartum)

SECONDARY OUTCOMES:
Functioning (measured at Weeks 24 and 52 postpartum)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Wisner, MD, Principal Investigator — Department of Psychiatry, University of Pittsburgh Medical Center
Locations (1):
- Women's Behavioral HealthCare Program, Pittsburgh, Pennsylvania, United States